CLINICAL TRIAL: NCT02818231
Title: Mechanisms of Cancerogenesis for Woodworkers Adenocarcinomas: Transcriptional Study of Olfactory Cleft Cells of Patients Exposed or Not to Wood Dust
Brief Title: Mechanisms of Cancerogenesis of Woodworkers Adenocarcinomas
Acronym: ADK-FO
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-A02004-45
Record Dates: First submitted 2016-05-23; First posted 2016-06-29 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2016-06

CONDITIONS: Ethmoid Sinus Adenocarcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — olfactory mucosae cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NON EXPOSED: Male, >50 years, unexposed to wood dust, without any nasal pathology, without known tumor
  -> Brushing of the olfactory cleft
  Interventions: Other: Brushing of the olfactory cleft
- EXPOSED: Male, >50 years, exposed to wood dust, without any nasal pathology, without known tumor
  -> Brushing of the olfactory cleft
  Interventions: Other: Brushing of the olfactory cleft

INTERVENTIONS:
Other: Brushing of the olfactory cleft — Non invasive sampling of olfactory cleft cells, by brushing under local anesthesia during fiberendoscopy Form: survey of acceptability

SUMMARY:
Nasal adenocarcinomas are closely related to wood dust exposure. The precise mechanisms of carcinogenesis leading to the transformation of the respiratory mucosa into a colonic-like mucosa remain unknown: chronic exposure to wood dust may cause chronic inflammation that may lead to pre-degenerative lesions, hypothesis yet unconfirmed. The tumor development requires the activation of a particular gene: CDX2. The working hypothesis is that chronic wood dust exposure is responsible for changes in genes of inflammation, which can in turn lead to changes in the expression of CDX2 and its cofactors, thus making possible the genesis of adenocarcinoma. This work is a pilot study aiming to better understand the mechanisms of carcinogenesis, and to study the feasibility of a larger prospective screening for woodworkers adenocarcinomas. Cells will be obtained from the at risk area (olfactory cleft) by a noninvasive method (brushing) in healthy volunteers (unexposed to wood dust) and in exposed volunteers to compare their genomes and study the genomic changes related to wood dust exposure.

DETAILED DESCRIPTION:
Pilot study, single center, prospective and retrospective, aiming to better understand the mechanisms of carcinogenesis of nasal adenocarcinoma among 2 groups of subjects based on their potential risk of nasal adenocarcinoma.

Patients will be recruited prospectively, in the ENT department (Prof. R. JANKOWSKI-Institut Lorrain Heart and vessels Louis Mathieu -Hospitals Brabois-CHU Nancy), during a visit for another medical reason.

They will be divided into 2 groups as follows:

* Group 1: NON EXPOSED : control group: patients not exposed to wood dust (low risk)
* Group 2: EXPOSED: patients exposed to wood dust (high risk)

After complete information, inclusion in the study will be proposed to patients

If inclusion is accepted, patients will undergo, during the nasal fiber endoscopy (performed for care), and under local anesthesia (performed for care), a brushing of the most accessible olfactory clef (performed for research). These samples will be compared to tumor samples which are already available (REFCOR)

The samples of groups 1 and 2 will be sent directly to the laboratory of Pathological Anatomy Cytology (Pr-J.M. VIGNAUD Hospital Brabois- CHU Nancy). They will briefly vortexed (5 min) and frozen. They will be kept in the laboratory of Pathological Anatomy Cytology (Pr-J.M. VIGNAUD Hospital Brabois- CHU Nancy) until analysis. The samples will be transferred from the laboratory of Pathological Anatomy Cytology (Pr-J.M. VIGNAUD Hospital Brabois- CHU Nancy) to the Genomics Platform (INSERM, U954, Prof. JL GUEANT- Faculty of Medicine, University of Lorraine), for analysis.

RNA will be extracted from olfactory cells , using RNeasy Mini kit (Qiagen) with DNase treatment. The concentration and purity of the DNA / RNA will be measured (OD at 230nm, 260nm and 280nm) with a Nanodrop spectrophotometer (Nyxor). The RNA integrity will be determined from the profiles of ribosomal RNAs (18S & 28S) measured on LabOnChip® (2100 Bioanalyzer System, Agilent Technologies). The RNA samples will be stored at -80 ° C until use.

The transcriptome analysis will be conducted on chips Whole Human Genome 60K * 8 developed by Agilent®, and according to the manufacturer's protocol (single-color Agilent protocol).

At the end of the research samples will be destroyed.

ELIGIBILITY:
Inclusion Criteria:

* Male, > 50 years
* No known tumor
* patient needing fiberendoscopy, but for nasal pathology
* informed consent given
* affiliation to a healthcare scheme compulsory
* prior medical exam 'NON EXPOSED' group: no wood dust exposure 'EXPOSED' group : wood dust exposure > 20 years with delay since the beginning of exposure > 30 years

Exclusion criteria:

* Prior radiotherapy on sinus or nasal fossa
* Inflammatory disease of nasal fossa
* Genetic disease with cancer risk (xeroderma pigmentosum, chromosomal abnormality deletion or translocation, DNA repair deficiency)
* No informed consent
* No affiliation to a healthcare scheme compulsory
* prior medical exam
* Contra-indication to Xylocaine

Ages: 50 Years to 120 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consultation requiring fiberendoscopy, planned in the ENT department of the CHRU of Nancy, in a context of routine care or of monitoring of professionnal wood dust exposure
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2016-06; Primary Completion 2016-09 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
The identification of expression profiles specific of wood dust exposure (comparison of both groups (exposed / non exposed)) | through study completion, an average of 1 year
  Descriptive data (Mean, Median, Min, Max). Comparison of gene expression levels ( Ttest ) of both groups: identification of expression profiles specific of each group (Ftest)

SECONDARY OUTCOMES:
The identification of expression profiles predictive of a nasal adenocarcinoma transformation. | through study completion, an average of 1 year
  Comparison of gene expression levels of the 15 exposed patients with known gene expression levels of 15 tumor samples (intestinal adenocarcinomas related to wood dust) (T Test) Identification of common modifications of gene expression (Ftest)
The acceptability of the brushing technique | through study completion, an average of 1 year
  The acceptability will be evaluated on a composite criterion with three sub-criteria
  * subjective representation of the utility of the screening (mean >5/10)
  * subjective evaluation of the acceptability (pain, discomfort, complication) (mean>5/10)
  * agreement for an eventual second sample (>90%) All sub-criteria must be fulfilled to meet this outcome

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Gallet, MD, Principal Investigator — CHRU Nancy
Locations (1):
- Service ORL-CHRU NANCY, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No